CLINICAL TRIAL: NCT02735824
Title: Genetic Study of Immunodeficiency: Search for New Genetic Causes for Primary Immunodeficiencies
Acronym: GSI
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University Children's Hospital Basel (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: GSI KEK_2015-0555
Record Dates: First submitted 2016-03-10; First posted 2016-04-13 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Immunologic Deficiency Syndromes
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA PBMC
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with suspected PID: From included patients with suspected primary immunodeficiency (PID), i.e. patients with recurrent/unusual infection, immune dysregulation and/or susceptibility to malignancies from whom consent to participate was obtained, nucleated blood cells and/or fibroblasts from skin biopsy will be used for genetic testing and functional assays. Blood serum will be used for antibody and cytokine measurement.
  Interventions: Procedure: blood sampling and skin biopsy
- healthy relatives of patients with PID: From healthy relatives of patients with suspected PID from whom consent to participate was obtained, nucleated cells will be used for genetic testing in order to compare their genetic information with the one form their relatives with suspected PID.
  Interventions: Procedure: blood sampling or mouth swap
- Healthy volunteers: From healthy volunteers from whom consent to participate was obtained, nucleated blood cells will be used for genetic testing and functional assays. Blood serum will be used for antibody and cytokine measurement. The data obtained will be compared to age matched patients with suspected PID.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling and skin biopsy — Nucleated blood cells and/or fibroblasts from skin biopsy will be used for genetic testing and functional assays. Blood serum will be used for antibody and cytokine measurement.
  Groups: patients with suspected PID
Procedure: blood sampling or mouth swap — specimen will be used for genetic testing, results compared to patients
  Groups: healthy relatives of patients with PID
Procedure: blood sampling — Nucleated blood cells and/or fibroblasts from skin biopsy will be used for genetic testing and functional assays. Blood serum will be used for antibody and cytokine measurement.
  Groups: Healthy volunteers

SUMMARY:
Individuals with suspected primary immunodeficiency will be studied and the results compared with healthy controls. Primary immunodeficiency may manifest as recurrent, severe or unusual infections as well as signs and symptoms of immune dysregulation such as autoimmunity or lymphoproliferation.

DETAILED DESCRIPTION:
Patients with a suspected immunodeficiency will be identified and invited to participate. Upon agreement, an additional blood sample will be collected when they have their routine bloods taken. If the study participants undergoes anaesthesia for any other reason, a small skin biopsy will be taken as well. Additional samples including blood samples or mouth swabs will be taken from healthy family members. Blood from healthy controls will only be taken when there is a clinical need for blood sampling (or when the study participant is already anaesthetised for any other reason) and not for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Patient with suspected PID, healthy relative or healthy volunteer
* consent

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: population from which the groups or cohorts will be selected: in- and outpatient clinic of the Division of Immunology, Univ. Chlindren's Hospital zurich
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-02; Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with suspected PID for whom a genetic cause has been identified | Through study completion, an average of 3 years
  Number of patients with suspected primary immunodeficiency included in the study for whom a diagnosis can be made with the genetic and functional data obtained from patients, their relatives and healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Jana M Pachlopnik Schmid, MD PhD, Principal Investigator — University Children's Hospital, Zurich
Locations (2):
- Switzerland (2):
  - Division of Immunology, Zurich, Canton of Zurich
  - University of Basel Children's Hospital, Basel

IPD SHARING:
Plan to Share IPD: Yes
planned publication in peer reviewed journals (PubMed)

REFERENCES:
- [Background] Vavassori S, Galson JD, Truck J, van den Berg A, Tamminga RYJ, Magerus-Chatinet A, Pelle O, Camenisch Gross U, Marques Maggio E, Prader S, Opitz L, Nuesch U, Mauracher A, Volkmer B, Speer O, Suda L, Rothlisberger B, Zimmermann DR, Muller R, Diepstra A, Visser L, Haralambieva E, Neven B, Rieux-Laucat F, Pachlopnik Schmid J. Lymphadenopathy driven by TCR-Vgamma8Vdelta1 T-cell expansion in FAS-related autoimmune lymphoproliferative syndrome. Blood Adv. 2017 Jun 22;1(15):1101-1106. doi: 10.1182/bloodadvances.2017006411. eCollection 2017 Jun 27. PMID 29296752
- [Background] Lewandowska DW, Capaul R, Prader S, Zagordi O, Geissberger FD, Kugler M, Knorr M, Berger C, Gungor T, Reichenbach J, Shah C, Boni J, Zbinden A, Trkola A, Pachlopnik Schmid J, Huber M. Persistent mammalian orthoreovirus, coxsackievirus and adenovirus co-infection in a child with a primary immunodeficiency detected by metagenomic sequencing: a case report. BMC Infect Dis. 2018 Jan 11;18(1):33. doi: 10.1186/s12879-018-2946-7. PMID 29325543
- [Background] Simonis A, Fux M, Nair G, Mueller NJ, Haralambieva E, Pabst T, Pachlopnik Schmid J, Schmidt A, Schanz U, Manz MG, Muller AMS. Allogeneic hematopoietic cell transplantation in patients with GATA2 deficiency-a case report and comprehensive review of the literature. Ann Hematol. 2018 Oct;97(10):1961-1973. doi: 10.1007/s00277-018-3388-4. Epub 2018 Jun 13. PMID 29947977
- [Background] Mauracher AA, Gujer E, Bachmann LM, Gusewell S, Pachlopnik Schmid J. Patterns of Immune Dysregulation in Primary Immunodeficiencies: A Systematic Review. J Allergy Clin Immunol Pract. 2021 Feb;9(2):792-802.e10. doi: 10.1016/j.jaip.2020.10.057. Epub 2020 Nov 11. PMID 33186766
- [Background] Truck J, Prader S, Natalucci G, Hagmann C, Brotschi B, Kelly J, Bassler D, Steindl K, Rauch A, Baumgartner M, Fingerhut R, Hauri-Hohl M, Gungor T, Pachlopnik Schmid J, Berger C, Reichenbach J. Swiss newborn screening for severe T and B cell deficiency with a combined TREC/KREC assay - management recommendations. Swiss Med Wkly. 2020 Jun 24;150:w20254. doi: 10.4414/smw.2020.20254. eCollection 2020 Jun 15. PMID 32579701
- [Background] Mauracher AA, Pagliarulo F, Faes L, Vavassori S, Gungor T, Bachmann LM, Pachlopnik Schmid J. Causes of low neonatal T-cell receptor excision circles: A systematic review. J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1457-1460.e22. doi: 10.1016/j.jaip.2017.02.009. Epub 2017 Mar 27. No abstract available. PMID 28359806
- [Background] Lemoine R, Pachlopnik-Schmid J, Farin HF, Bigorgne A, Debre M, Sepulveda F, Heritier S, Lemale J, Talbotec C, Rieux-Laucat F, Ruemmele F, Morali A, Cathebras P, Nitschke P, Bole-Feysot C, Blanche S, Brousse N, Picard C, Clevers H, Fischer A, de Saint Basile G. Immune deficiency-related enteropathy-lymphocytopenia-alopecia syndrome results from tetratricopeptide repeat domain 7A deficiency. J Allergy Clin Immunol. 2014 Dec;134(6):1354-1364.e6. doi: 10.1016/j.jaci.2014.07.019. Epub 2014 Aug 28. PMID 25174867
- [Background] Pachlopnik Schmid J, Gungor T, Seger R. Modern management of primary T-cell immunodeficiencies. Pediatr Allergy Immunol. 2014 Jun;25(4):300-13. doi: 10.1111/pai.12179. Epub 2014 Jan 3. PMID 24383740
- [Background] Planas R, Felber M, Vavassori S, Pachlopnik Schmid J. The hyperinflammatory spectrum: from defects in cytotoxicity to cytokine control. Front Immunol. 2023 Apr 28;14:1163316. doi: 10.3389/fimmu.2023.1163316. eCollection 2023. PMID 37187762
- [Background] Prader S, Ritz N, Baleydier F, Andre MC, Stahli N, Schmid K, Schmid H, Woerner A, Diesch T, Meyer Sauteur PM, Truck J, Gebistorf F, Opitz L, Killian MP, Marchetti T, Vavassori S, Blanchard-Rohner G, Mc Lin V, Grazioli S, Pachlopnik Schmid J. X-Linked Lymphoproliferative Disease Mimicking Multisystem Inflammatory Syndrome in Children-A Case Report. Front Pediatr. 2021 Aug 3;9:691024. doi: 10.3389/fped.2021.691024. eCollection 2021. PMID 34414143
- [Background] Vavassori S, Chou J, Faletti LE, Haunerdinger V, Opitz L, Joset P, Fraser CJ, Prader S, Gao X, Schuch LA, Wagner M, Hoefele J, Maccari ME, Zhu Y, Elakis G, Gabbett MT, Forstner M, Omran H, Kaiser T, Kessler C, Olbrich H, Frosk P, Almutairi A, Platt CD, Elkins M, Weeks S, Rubin T, Planas R, Marchetti T, Koovely D, Klambt V, Soliman NA, von Hardenberg S, Klemann C, Baumann U, Lenz D, Klein-Franke A, Schwemmle M, Huber M, Sturm E, Hartleif S, Haffner K, Gimpel C, Brotschi B, Laube G, Gungor T, Buckley MF, Kottke R, Staufner C, Hildebrandt F, Reu-Hofer S, Moll S, Weber A, Kaur H, Ehl S, Hiller S, Geha R, Roscioli T, Griese M, Pachlopnik Schmid J. Multisystem inflammation and susceptibility to viral infections in human ZNFX1 deficiency. J Allergy Clin Immunol. 2021 Aug;148(2):381-393. doi: 10.1016/j.jaci.2021.03.045. Epub 2021 Apr 17. PMID 33872655
- [Result] Marquardt L, Lacour M, Hoernes M, Opitz L, Lecca R, Volkmer B, Reichenbach J, Hohl D, Ansari M, Ozsahin H, Gungor T, Pachlopnik Schmid J. Unusual dermatological presentation and immune phenotype in SCID due to an IL7R mutation: the value of whole-exome sequencing and the potential benefit of newborn screening. J Eur Acad Dermatol Venereol. 2017 Mar;31(3):e147-e148. doi: 10.1111/jdv.13888. Epub 2016 Sep 5. No abstract available. PMID 27593400
- [Result] Schwab C, Gabrysch A, Olbrich P, Patino V, Warnatz K, Wolff D, Hoshino A, Kobayashi M, Imai K, Takagi M, Dybedal I, Haddock JA, Sansom DM, Lucena JM, Seidl M, Schmitt-Graeff A, Reiser V, Emmerich F, Frede N, Bulashevska A, Salzer U, Schubert D, Hayakawa S, Okada S, Kanariou M, Kucuk ZY, Chapdelaine H, Petruzelkova L, Sumnik Z, Sediva A, Slatter M, Arkwright PD, Cant A, Lorenz HM, Giese T, Lougaris V, Plebani A, Price C, Sullivan KE, Moutschen M, Litzman J, Freiberger T, van de Veerdonk FL, Recher M, Albert MH, Hauck F, Seneviratne S, Pachlopnik Schmid J, Kolios A, Unglik G, Klemann C, Speckmann C, Ehl S, Leichtner A, Blumberg R, Franke A, Snapper S, Zeissig S, Cunningham-Rundles C, Giulino-Roth L, Elemento O, Duckers G, Niehues T, Fronkova E, Kanderova V, Platt CD, Chou J, Chatila TA, Geha R, McDermott E, Bunn S, Kurzai M, Schulz A, Alsina L, Casals F, Deya-Martinez A, Hambleton S, Kanegane H, Tasken K, Neth O, Grimbacher B. Phenotype, penetrance, and treatment of 133 cytotoxic T-lymphocyte antigen 4-insufficient subjects. J Allergy Clin Immunol. 2018 Dec;142(6):1932-1946. doi: 10.1016/j.jaci.2018.02.055. Epub 2018 May 4. PMID 29729943
- [Result] Maccari ME, Abolhassani H, Aghamohammadi A, Aiuti A, Aleinikova O, Bangs C, Baris S, Barzaghi F, Baxendale H, Buckland M, Burns SO, Cancrini C, Cant A, Cathebras P, Cavazzana M, Chandra A, Conti F, Coulter T, Devlin LA, Edgar JDM, Faust S, Fischer A, Garcia-Prat M, Hammarstrom L, Heeg M, Jolles S, Karakoc-Aydiner E, Kindle G, Kiykim A, Kumararatne D, Grimbacher B, Longhurst H, Mahlaoui N, Milota T, Moreira F, Moshous D, Mukhina A, Neth O, Neven B, Nieters A, Olbrich P, Ozen A, Pachlopnik Schmid J, Picard C, Prader S, Rae W, Reichenbach J, Rusch S, Savic S, Scarselli A, Scheible R, Sediva A, Sharapova SO, Shcherbina A, Slatter M, Soler-Palacin P, Stanislas A, Suarez F, Tucci F, Uhlmann A, van Montfrans J, Warnatz K, Williams AP, Wood P, Kracker S, Condliffe AM, Ehl S. Disease Evolution and Response to Rapamycin in Activated Phosphoinositide 3-Kinase delta Syndrome: The European Society for Immunodeficiencies-Activated Phosphoinositide 3-Kinase delta Syndrome Registry. Front Immunol. 2018 Mar 16;9:543. doi: 10.3389/fimmu.2018.00543. eCollection 2018. PMID 29599784
- [Result] Meshaal SS, El Hawary RE, Abd Elaziz DS, Eldash A, Alkady R, Lotfy S, Mauracher AA, Opitz L, Pachlopnik Schmid J, van der Burg M, Chou J, Galal NM, Boutros JA, Geha R, Elmarsafy AM. Phenotypical heterogeneity in RAG-deficient patients from a highly consanguineous population. Clin Exp Immunol. 2019 Feb;195(2):202-212. doi: 10.1111/cei.13222. Epub 2018 Nov 4. PMID 30307608
- [Result] El Hawary RE, Mauracher AA, Meshaal SS, Eldash A, Abd Elaziz DS, Alkady R, Lotfy S, Opitz L, Galal NM, Boutros JA, Pachlopnik Schmid J, Elmarsafy AM. MHC-II Deficiency Among Egyptians: Novel Mutations and Unique Phenotypes. J Allergy Clin Immunol Pract. 2019 Mar;7(3):856-863. doi: 10.1016/j.jaip.2018.07.046. Epub 2018 Aug 28. PMID 30170160
- [Result] Prader S, Felber M, Volkmer B, Truck J, Schwieger-Briel A, Theiler M, Weibel L, Hambleton S, Seipel K, Vavassori S, Pachlopnik Schmid J. Life-Threatening Primary Varicella Zoster Virus Infection With Hemophagocytic Lymphohistiocytosis-Like Disease in GATA2 Haploinsufficiency Accompanied by Expansion of Double Negative T-Lymphocytes. Front Immunol. 2018 Dec 3;9:2766. doi: 10.3389/fimmu.2018.02766. eCollection 2018. PMID 30564229
- [Result] Volkmer B, Planas R, Gossweiler E, Lunemann A, Opitz L, Mauracher A, Nuesch U, Gayden T, Kaiser D, Drexel B, Dumrese C, Jabado N, Vavassori S, Pachlopnik Schmid J. Recurrent inflammatory disease caused by a heterozygous mutation in CD48. J Allergy Clin Immunol. 2019 Nov;144(5):1441-1445.e17. doi: 10.1016/j.jaci.2019.07.038. Epub 2019 Aug 13. No abstract available. PMID 31419545
- [Result] Mauracher AA, Eekels JJM, Woytschak J, van Drogen A, Bosch A, Prader S, Felber M, Heeg M, Opitz L, Truck J, Schroeder S, Adank E, Klocperk A, Haralambieva E, Zimmermann D, Tantou S, Kotsonis K, Stergiou A, Kanariou MG, Ehl S, Boyman O, Sediva A, Renella R, Schmugge M, Vavassori S, Pachlopnik Schmid J. Erythropoiesis defect observed in STAT3 GOF patients with severe anemia. J Allergy Clin Immunol. 2020 Apr;145(4):1297-1301. doi: 10.1016/j.jaci.2019.11.042. Epub 2019 Dec 17. No abstract available. PMID 31857100
- [Result] Ghraichy M, Galson JD, Kovaltsuk A, von Niederhausern V, Pachlopnik Schmid J, Recher M, Jauch AJ, Miho E, Kelly DF, Deane CM, Truck J. Maturation of the Human Immunoglobulin Heavy Chain Repertoire With Age. Front Immunol. 2020 Aug 6;11:1734. doi: 10.3389/fimmu.2020.01734. eCollection 2020. PMID 32849618
- [Result] El Hawary R, Meshaal S, Mauracher AA, Opitz L, Abd Elaziz D, Lotfy S, Eldash A, Boutros J, Galal N, Pachlopnik Schmid J, Elmarsafy A. Whole-exome sequencing of T- B+ severe combined immunodeficiency in Egyptian infants, JAK3 predominance and novel variants. Clin Exp Immunol. 2021 Mar;203(3):448-457. doi: 10.1111/cei.13536. Epub 2020 Nov 2. PMID 33040328
- [Result] Fouriki A, Schnider C, Theodoropoulou K, Pachlopnik J, Hofer M, Candotti F. [Newborn screening for severe T and B lymphocyte deficiencies in Switzerland]. Rev Med Suisse. 2021 Jan 13;17(720-1):68-76. French. PMID 33443835
- [Result] Hanitsch L, Baumann U, Boztug K, Burkhard-Meier U, Fasshauer M, Habermehl P, Hauck F, Klock G, Liese J, Meyer O, Muller R, Pachlopnik-Schmid J, Pfeiffer-Kascha D, Warnatz K, Wehr C, Wittke K, Niehues T, von Bernuth H. Treatment and management of primary antibody deficiency: German interdisciplinary evidence-based consensus guideline. Eur J Immunol. 2020 Oct;50(10):1432-1446. doi: 10.1002/eji.202048713. Epub 2020 Sep 9. PMID 32845010
- [Result] Jagle S, Heeg M, Grun S, Rensing-Ehl A, Maccari ME, Klemann C, Jones N, Lehmberg K, Bettoni C, Warnatz K, Grimbacher B, Biebl A, Schauer U, Hague R, Neth O, Mauracher A, Pachlopnik Schmid J, Fabre A, Kostyuchenko L, Fuhrer M, Lorenz MR, Schwarz K, Rohr J, Ehl S. Distinct molecular response patterns of activating STAT3 mutations associate with penetrance of lymphoproliferation and autoimmunity. Clin Immunol. 2020 Jan;210:108316. doi: 10.1016/j.clim.2019.108316. Epub 2019 Nov 23. PMID 31770611
- [Result] Grazioli S, Tavaglione F, Torriani G, Wagner N, Rohr M, L'Huillier AG, Leclercq C, Perrin A, Bordessoule A, Beghetti M, Schmid JP, Vavassori S, Perreau M, Eberhardt C, Didierlaurent A, Kaiser L, Eckerle I, Roux-Lombard P, Blanchard-Rohner G. Immunological Assessment of Pediatric Multisystem Inflammatory Syndrome Related to Coronavirus Disease 2019. J Pediatric Infect Dis Soc. 2021 Aug 14;10(6):706-713. doi: 10.1093/jpids/piaa142. PMID 33180935
- [Result] Blanchard-Rohner G, Pachlopnik Schmid J, Candotti F, Hofer M. [Pediatric COVID-19 - Pathophysiology, immune responses, genetic predispositions, hyperinflammatory syndrome]. Rev Med Suisse. 2021 Feb 17;17(726):334-337. French. PMID 33599408
- [Result] Fouriki A, Fougere Y, De Camaret C, Blanchard Rohner G, Grazioli S, Wagner N, Relly C, Pachlopnik Schmid J, Truck J, Kottanatu L, Perez E, Perez MH, Schaffner D, Asner SA, Hofer M. Case Report: Case Series of Children With Multisystem Inflammatory Syndrome Following SARS-CoV-2 Infection in Switzerland. Front Pediatr. 2021 Jan 5;8:594127. doi: 10.3389/fped.2020.594127. eCollection 2020. PMID 33469522
- [Result] Dedual MA, Wueest S, Challa TD, Lucchini FC, Aeppli TRJ, Borsigova M, Mauracher AA, Vavassori S, Pachlopnik Schmid J, Bluher M, Konrad D. Obesity-Induced Increase in Cystatin C Alleviates Tissue Inflammation. Diabetes. 2020 Sep;69(9):1927-1935. doi: 10.2337/db19-1206. Epub 2020 Jul 2. PMID 32616516
- [Result] Felber M, Steward CG, Kentouche K, Fasth A, Wynn RF, Zeilhofer U, Haunerdinger V, Volkmer B, Prader S, Gruhn B, Ehl S, Lehmberg K, Muller D, Gennery AR, Albert MH, Hauck F, Rao K, Veys P, Hassan M, Lankester AC, Schmid JP, Hauri-Hohl MM, Gungor T. Targeted busulfan-based reduced-intensity conditioning and HLA-matched HSCT cure hemophagocytic lymphohistiocytosis. Blood Adv. 2020 May 12;4(9):1998-2010. doi: 10.1182/bloodadvances.2020001748. PMID 32384542
- [Result] Weins AB, Theiler M, Bogatu B, Kerl K, Pleimes M, Pachlopnik-Schmid J, Weibel L. Febrile ulceronecrotic Mucha-Habermann disease mimicking Kawasaki disease. J Dtsch Dermatol Ges. 2020 Feb;18(2):140-142. doi: 10.1111/ddg.13989. Epub 2019 Dec 9. No abstract available. PMID 31814284
- [Result] Nuesch U, Mauracher AA, Opitz L, Volkmer B, Michalak-Micka K, Kamarashev J, Hartwig T, Reichmann E, Becher B, Vavassori S, Pachlopnik Schmid J. Epithelial proliferation in inflammatory skin disease is regulated by tetratricopeptide repeat domain 7 (Ttc7) in fibroblasts and lymphocytes. J Allergy Clin Immunol. 2019 Jan;143(1):292-304.e8. doi: 10.1016/j.jaci.2018.02.057. Epub 2018 Jun 14. PMID 29775636
- [Result] Giannelou A, Wang H, Zhou Q, Park YH, Abu-Asab MS, Ylaya K, Stone DL, Sediva A, Sleiman R, Sramkova L, Bhatla D, Serti E, Tsai WL, Yang D, Bishop K, Carrington B, Pei W, Deuitch N, Brooks S, Edwan JH, Joshi S, Prader S, Kaiser D, Owen WC, Sonbul AA, Zhang Y, Niemela JE, Burgess SM, Boehm M, Rehermann B, Chae J, Quezado MM, Ombrello AK, Buckley RH, Grom AA, Remmers EF, Pachlopnik JM, Su HC, Gutierrez-Cruz G, Hewitt SM, Sood R, Risma K, Calvo KR, Rosenzweig SD, Gadina M, Hafner M, Sun HW, Kastner DL, Aksentijevich I. Aberrant tRNA processing causes an autoinflammatory syndrome responsive to TNF inhibitors. Ann Rheum Dis. 2018 Apr;77(4):612-619. doi: 10.1136/annrheumdis-2017-212401. Epub 2018 Jan 22. PMID 29358286
- [Result] Schepp J, Proietti M, Frede N, Buchta M, Hubscher K, Rojas Restrepo J, Goldacker S, Warnatz K, Pachlopnik Schmid J, Duppenthaler A, Lougaris V, Uriarte I, Kelly S, Hershfield M, Grimbacher B. Screening of 181 Patients With Antibody Deficiency for Deficiency of Adenosine Deaminase 2 Sheds New Light on the Disease in Adulthood. Arthritis Rheumatol. 2017 Aug;69(8):1689-1700. doi: 10.1002/art.40147. Epub 2017 Jul 5. PMID 28493328
- [Result] Miot C, Imai K, Imai C, Mancini AJ, Kucuk ZY, Kawai T, Nishikomori R, Ito E, Pellier I, Dupuis Girod S, Rosain J, Sasaki S, Chandrakasan S, Pachlopnik Schmid J, Okano T, Colin E, Olaya-Vargas A, Yamazaki-Nakashimada M, Qasim W, Espinosa Padilla S, Jones A, Krol A, Cole N, Jolles S, Bleesing J, Vraetz T, Gennery AR, Abinun M, Gungor T, Costa-Carvalho B, Condino-Neto A, Veys P, Holland SM, Uzel G, Moshous D, Neven B, Blanche S, Ehl S, Doffinger R, Patel SY, Puel A, Bustamante J, Gelfand EW, Casanova JL, Orange JS, Picard C. Hematopoietic stem cell transplantation in 29 patients hemizygous for hypomorphic IKBKG/NEMO mutations. Blood. 2017 Sep 21;130(12):1456-1467. doi: 10.1182/blood-2017-03-771600. Epub 2017 Jul 5. PMID 28679735
- [Result] Ter Haar NM, Jeyaratnam J, Lachmann HJ, Simon A, Brogan PA, Doglio M, Cattalini M, Anton J, Modesto C, Quartier P, Hoppenreijs E, Martino S, Insalaco A, Cantarini L, Lepore L, Alessio M, Calvo Penades I, Boros C, Consolini R, Rigante D, Russo R, Pachlopnik Schmid J, Lane T, Martini A, Ruperto N, Frenkel J, Gattorno M; Paediatric Rheumatology International Trials Organisation and Eurofever Project. The Phenotype and Genotype of Mevalonate Kinase Deficiency: A Series of 114 Cases From the Eurofever Registry. Arthritis Rheumatol. 2016 Nov;68(11):2795-2805. doi: 10.1002/art.39763. PMID 27213830
- [Result] Ravelli A, Minoia F, Davi S, Horne A, Bovis F, Pistorio A, Arico M, Avcin T, Behrens EM, De Benedetti F, Filipovic L, Grom AA, Henter JI, Ilowite NT, Jordan MB, Khubchandani R, Kitoh T, Lehmberg K, Lovell DJ, Miettunen P, Nichols KE, Ozen S, Pachlopnik Schmid J, Ramanan AV, Russo R, Schneider R, Sterba G, Uziel Y, Wallace C, Wouters C, Wulffraat N, Demirkaya E, Brunner HI, Martini A, Ruperto N, Cron RQ; Paediatric Rheumatology International Trials Organisation; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology Collaborative Study Group; Histiocyte Society. 2016 Classification Criteria for Macrophage Activation Syndrome Complicating Systemic Juvenile Idiopathic Arthritis: A European League Against Rheumatism/American College of Rheumatology/Paediatric Rheumatology International Trials Organisation Collaborative Initiative. Ann Rheum Dis. 2016 Mar;75(3):481-9. doi: 10.1136/annrheumdis-2015-208982. PMID 26865703
- [Result] Bode SF, Ammann S, Al-Herz W, Bataneant M, Dvorak CC, Gehring S, Gennery A, Gilmour KC, Gonzalez-Granado LI, Gross-Wieltsch U, Ifversen M, Lingman-Framme J, Matthes-Martin S, Mesters R, Meyts I, van Montfrans JM, Pachlopnik Schmid J, Pai SY, Soler-Palacin P, Schuermann U, Schuster V, Seidel MG, Speckmann C, Stepensky P, Sykora KW, Tesi B, Vraetz T, Waruiru C, Bryceson YT, Moshous D, Lehmberg K, Jordan MB, Ehl S; Inborn Errors Working Party of the EBMT. The syndrome of hemophagocytic lymphohistiocytosis in primary immunodeficiencies: implications for differential diagnosis and pathogenesis. Haematologica. 2015 Jul;100(7):978-88. doi: 10.3324/haematol.2014.121608. Epub 2015 May 28. PMID 26022711
- [Result] Sepulveda FE, Debeurme F, Menasche G, Kurowska M, Cote M, Pachlopnik Schmid J, Fischer A, de Saint Basile G. Distinct severity of HLH in both human and murine mutants with complete loss of cytotoxic effector PRF1, RAB27A, and STX11. Blood. 2013 Jan 24;121(4):595-603. doi: 10.1182/blood-2012-07-440339. Epub 2012 Nov 16. PMID 23160464
- [Derived] Kannan A, Suomalainen M, Volle R, Bauer M, Amsler M, Trinh HV, Vavassori S, Schmid JP, Vilhena G, Marin-Gonzalez A, Perez R, Franceschini A, Mering CV, Hemmi S, Greber UF. Sequence-Specific Features of Short Double-Strand, Blunt-End RNAs Have RIG-I- and Type 1 Interferon-Dependent or -Independent Anti-Viral Effects. Viruses. 2022 Jun 28;14(7):1407. doi: 10.3390/v14071407. PMID 35891387